CLINICAL TRIAL: NCT07023939
Title: Comparative Study on the Clinical Outcomes of Restoring Dentine Caries Lesions in Primary Molars Using Silver Modified Versus Conventional Atraumatic Restorative Treatment (A Randomized Clinical Trial)
Brief Title: Atraumatic Versus Silver-Modified Atraumatic Restorative Treatment in Primary Molars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beirut Arab University (Other)
Responsible Party: Principal Investigator, Sana Solh, Clinical Instructor, Beirut Arab University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-H-011-D-M-0489
Record Dates: First submitted 2025-05-23; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Dental Caries; Dental Caries in Children
Keywords: Early Childhood caries; SilverDiamine flouride; Glass Ionomer Cement; Minimal Intervention Dentistry
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: split mouth design
Who Masked: Participant
Masking Description: The data analyst performing statistical evaluations was masked to group allocation during the initial analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ART- Atraumatic Restorative Treatment (Active Comparator): Children received Atraumatic Restorative Treatment (ART), which involved selective caries removal using hand instruments and restoration with high-viscosity glass ionomer cement. Carious dentin was excavated from the axial walls with a spoon excavator, unsupported enamel was removed with a hatchet, and only soft demineralized dentin on the pulpal floor was removed until firm dentin was reached.
  Interventions: Drug: ART: Atraumatic restorative treatment, SMART: Silver-Modified Atraumatic Restorative Treatment
- SMART_Silver-Modified Atraumatic Restorative Treatment (Experimental): Children received Silver-Modified Atraumatic Restorative Treatment (SMART), which included the application of 38% silver diamine fluoride (SDF) followed by ART. Gingival tissues and lips were protected with petroleum jelly. One drop of SDF (Advantage Arrest™, Elevate Oral Care, USA) was placed into a disposable dish and applied to affected tooth surfaces using a bent micro-sponge for at least 60 seconds. Excess was blotted with a cotton pellet, and the area was air-dried under isolation for up to three minutes. ART was then completed using high-viscosity glass ionomer cement.
  Interventions: Drug: ART: Atraumatic restorative treatment, SMART: Silver-Modified Atraumatic Restorative Treatment

INTERVENTIONS:
Drug: ART: Atraumatic restorative treatment, SMART: Silver-Modified Atraumatic Restorative Treatment — ART Group:
  Selective caries removal was done using hand instruments-carious dentin was excavated from the axial walls with a spoon excavator, and unsupported enamel was carefully removed using a hatchet. On the pulpal floor, only soft, completely demineralized dentin was removed until firm dentin was reached.
  SMART Group:
  the surrounding gingival tissues and lips were protected with petroleum jelly to avoid staining and irritation (2) ) one drop of SDF (Advantage Arrest ™, Elevate Oral Care, USA) was placed into a disposable dish, (4) SDF was applied with a bended micro-sponge directly to the affected tooth surfaces for minimum of 60 seconds, (3) excess was blotted with a cotton pellet, (4)and the area was air-dried while maintaining isolation for up to three minutes.

SUMMARY:
The goal of this clinical trial is to evaluate and compare the short-term effectiveness of two minimally invasive treatments-Atraumatic Restorative Treatment (ART) and Silver-Modified Atraumatic Restorative Treatment (SMART)-in managing dentine caries lesions in the primary molars of children aged 3 to 7 years with Early Childhood Caries (ECC). The main questions it aims to answer are:

* Which treatment method (ART or SMART) results in higher clinical success after six months?
* How do ART and SMART treatments affect the Oral Health-Related Quality of Life (OHRQoL) of the children? The researcher will compare teeth restored using ART with those treated using SMART (which includes the application of silver diamine fluoride before restoration) to see if one approach leads to better restoration outcomes and to assess how these restorations will impact the quality of life.

Participants will:

* Receive both types of treatments in different teeth (split-mouth design).
* Undergo clinical evaluation of the treated teeth at baseline and six months to assess success based on restoration retention, integrity, and absence of secondary caries.
* Have their parents complete a quality-of-life questionnaire (A-ECOHIS) at the start and at the six-month follow-up.

DETAILED DESCRIPTION:
Aim of the Study in details:

Primary Aim

This study aims to evaluate and compare the clinical outcomes of Silver-Modified Atraumatic Restorative Treatment (SMART) and conventional Atraumatic Restorative Treatment (ART) in the management of carious primary molars in preschool children. This comparison includes:

* Success rate: which include restoration integrity, marginal adaptation, absence of secondary caries, and tooth vitality.
* Retention rate: Determined by monitoring whether the restoration remains fully or partially retained over time
* Caries arrest: where arrested lesions present with hard, darkened surfaces and no progression in lesion size Secondary Aim
* To describe the change in oral health-related quality of life of preschool children before and after placement of ART and SMART restorations Randomization The sample size was specified by using the G* power test, assuming a statistical level of significance of 95% and power of 80% with normal distribution, and effect size calculated from means and standard deviation of 2 groups obtained from a previous similar study (Jiang et al.,2021). The original sample size was 64 molars and was increased up to 80 to avoid any drop out.

Eligible molars were randomly and equally assigned to either the SMART or ART group using a randomization software (Random.org).

Calibration:

One calibrated examiner was responsible for all the dental examinations. The intra-examiner agreement was assessed by re-examining 10% of the sample. The Kappa statistic for intra-examiner reliability was 0.87 which indicates consistency in the application of scoring criteria over the study period.

Blinding and Outcome Assessment Follow up assessments were done by the operator at 6 months. Complete blinding was not feasible in some cases particularly where GIC restorations where lost due to noticeable staining of the cavity with SDF. However, blinding of the data analyst was done where all study data was labelled with non-identifying Alphabet letters to reduce risk of bias.

Data Collection:

At baseline, parents completed a two-part questionnaire: Part 1 gathered general demographic information, while Part 2 included the validated Arabic version of the Early Childhood Oral Health Impact Scale (A-ECOHIS) validated by Farsi et al in 2017[20]. At the second follow-up visit. parents completed the same questionnaire again.

Statistical Analysis Data were statistically analyzed through SPSS 28 (SPSS IBM statistics, USA). Based on the results of the Shapiro-Wilk test, most of the data were determined to follow a normal distribution. The significance level was set at p ≤ 0.05. Fishers exact test was used to compare the outcomes between ART and SMART at a single time point. Categorical data like the relation between the success rate of both treatments and the type of the cavity was analyzed by using the Chi-Square Test of Independence. Paired Samples t-Test was used to assess the changes in ECOHIS scores at baseline and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Study Participants: Generally healthy children aged 3 to 7 years
* Behavior Rating (Frankel's Scale):

Negative (Score 2) Positive (Score 3)

* Dental Condition: At least two bilateral asymptomatic decayed primary molars
* Caries Classification: based on International caries detection and assessment systemII I(CDAS II) Scores 4 & 5 (Occlusal or occluso-proximal carious dentin lesions)

Exclusion Criteria:

* Children with systemic diseases/conditions (ASA Type I)
* Behavior Rating (Frankel's Scale) Definitely positive(Score 1) Definitely negative (Score 4).
* Teeth showing irreversible pulpitis or pulpal pathology (abscess, fistula, mobility)
* Teeth with very deep cavities or score 6 based on ICDAS II

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
primary outcome : Success rate of restorations assessed by Modified ART Criteria | 6 months post-treatment
  The proportion of restorations that meet criteria for success based on Modified ART CRITERIA evaluation UNIT OF MEASURE: % OF restorations rated successful

SECONDARY OUTCOMES:
Change in Oral Health-Related Quality of Life (OHRQoL) assessed by Early Childhood Oral Health Impact Scale (ECOHIS) filled by parents | Baseline and 6-month follow-up
  Mean change in total ECOHIS score from baseline to 6 months post-treatment. The ECOHIS includes 13 items scored on a 5-point Likert scale (0 = never to 4 = very often). Total score range: 0-52. Higher scores indicate worse oral health-related quality of life.
  Unit of Measure: Mean score change on ECOHIS

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Ahmad Tarabaih, Assoc.Prof, Study Director — Department of Pediatric Dentistry, Beirut Arab university; Dr.Ahmad Holiel, Assis.Prof, Study Director — Department of Esthetic and Restorative Dentistry, Beirut Arab University
Locations (1):
- Beirut arab University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Solh SK, Holiel AA, Tarabaih AS. Atraumatic Versus Silver-Modified Atraumatic Restorative Treatment in Primary Molars: A Randomized Clinical Trial on Minimally Invasive Caries Management and Oral Health-Related Quality of Life. Clin Exp Dent Res. 2026 Feb;12(1):e70299. doi: 10.1002/cre2.70299. PMID 41632901

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/39/NCT07023939/Prot_SAP_ICF_000.pdf